CLINICAL TRIAL: NCT03547739
Title: Testing Strategies for Couple Engagement in PMTCT and Family Health in Kenya
Acronym: Jamii Bora
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Kenya Medical Research Institute (Other); University of Michigan (Other); University of Witwatersrand, South Africa (Other); University of Pennsylvania (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Janet M. Turan, PhD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300001427; 000518108 (Other: UAB Office of Sponsored Programs); R01MH116736 (NIH)
Record Dates: First submitted 2018-05-09; First posted 2018-06-06 (Actual); Results first posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-07

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — House Calls

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home visits (Active Comparator): Participants randomized to intervention arm receive 5 home visits conducted by one female and one male lay health worker.
  Interventions: Behavioral: Home visits
- HIV Self-testing (Active Comparator): Women in this study group will receive HIV self-test kits for themselves and their male partner at up to 4 time points.
  Interventions: Behavioral: HIV Self-testing
- Standard Care (No Intervention): Participants will receive current standard clinic-based services including the option for women and partners to return to the clinic for male partner HIV testing or Couples HIV Counseling and Testing (CHCT).

INTERVENTIONS:
Behavioral: Home visits — If a couple has been randomized to the home visit intervention arm, a lay health worker will obtain detailed locator information (including cell phone contacts) and consult with the couple about optimal times for a home visit. As described above, the intervention arm will consist of five home visits conducted by one female and one male lay health worker, including two home visits during pregnancy, one at six weeks after the birth, and two booster sessions, one at six months after the birth and one at 12 months after the birth. Home visits are designed for all pregnant couples (regardless of woman's initial HIV test result at the antenatal clinic) and include topics important for maternal, paternal, and child health during pregnancy and postpartum.
  Arms: Home visits
Behavioral: HIV Self-testing — Women in this study group will receive oral-fluid-based rapid HIV test kits for themselves and their male partner at up to 4 time points (twice during pregnancy and twice postpartum). Each test will be accompanied with a self-testing instruction sheet describing step-by-step procedures in multiple languages. Study staff will also conduct a brief demonstration on how to use the tests. Participants will be encouraged to offer a test kit to their male partner or to undertake couples testing. They will also be counseled on how to talk to their partners and the possibility of adverse partner reactions. Participants will be instructed to seek clinic-based confirmatory testing if a reactive self-test result is obtained.
  Arms: HIV Self-testing

SUMMARY:
This study will test the efficacy and cost-effectiveness of an interdependence theory-based couples intervention in Kenya that reaches pregnant women and male partners through home visits by male-female pairs of lay health workers, and includes offer of home-based CHTC services.

DETAILED DESCRIPTION:
Despite the potential for antiretroviral therapy to improve maternal health and reduce mother-to-child transmission of HIV to as low as 1%, HIV-related maternal deaths and HIV infection among infants remain unacceptably high across sub-Saharan Africa. This is particularly true in Kenya, where crucial drop-offs occur in the cascade of prevention of mother-to-child transmission (PMTCT) services. Weak health systems contribute to insufficient service coverage, but many barriers lie beyond the clinic-in the partner, family, and community factors that shape women's health decisions. The investigators' research in a high HIV prevalence area of southwestern Kenya has shown that many women avoid couples HIV testing and do not adhere to PMTCT regimens because they fear negative consequences from a male partner. Men can play a crucial supportive role for family health, but male partners in Kenya are poorly engaged in antenatal care and uptake of couples HIV testing during pregnancy is low. Pregnant women desire to be tested for HIV together with their partner and need the support for mutual disclosure involved in couples HIV testing and counseling (CHTC), regardless of whether they know their own HIV status. In this context, the investigators will test the efficacy of an interdependence theory-based couples intervention that reaches pregnant women and male partners through home visits by male-female pairs of lay health workers, and includes offer of home-based CHTC services. The randomized pilot study of this intervention with 96 pregnant couples (R34MH102103) demonstrated significant increases in uptake of couples testing (64% in intervention vs. 23% in control, p<0.001) and significant improvements in health behaviors such as exclusive breastfeeding and postpartum care. The investigators will now conduct a more robust investigation to determine whether this intervention improves uptake of couples HIV testing and health outcomes over and above less intensive male engagement strategies being used in the region. This theory-based couples intervention has strong potential to increase couple HIV testing and collaboration for family health. The study will inform decision-makers about cost-effective strategies to engage pregnant couples in PMTCT and family health, with important downstream benefits for maternal, paternal, and infant health.

ELIGIBILITY:
Inclusion Criteria:

* Women at 36 weeks of pregnancy or less
* 15 years of age or older
* Has been offered HIV testing at ANC
* Is currently in a stable relationship with a male partner and living with that male partner - Has not yet participated in couple HIV testing during this pregnancy.
* Male partner is the person identified by the pregnant woman as her primary male partner and should also be 15 years of age or older.
* Not in an HIV-positive concordant relationship.

Exclusion Criteria:

* Greater than 36 weeks of pregnancy
* Less than 15 years of age
* Not currently in a stable relationship with a male partner
* Does not currently live with male partner
* Has not been offered HIV testing at ANC

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet M Turan, PhD, MPH, Principal Investigator — University of Alabama at Birmingham; Lynae Darbes, PhD, Principal Investigator — University of Michigan
Locations (1):
- Kenya Medical Research Institute, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kwena Z, Kimbo L, Darbes LA, Hatcher AM, Helova A, Owino G, Thirumurthy H, Bukusi EA, Braun T, Kilgore M, Pisu M, Tamhane A, Nghiem VT, Agot K, Neilands TB, Turan JM. Testing strategies for couple engagement in prevention of mother-to-child transmission of HIV and family health in Kenya: study protocol for a randomized controlled trial. Trials. 2021 Jan 6;22(1):19. doi: 10.1186/s13063-020-04956-1. PMID 33407784
- [Result] Borgstede SJ, Elly A, Helova A, Kwena Z, Darbes LA, Hatcher A, Thirumurthy H, Owino G, Pisu M, Owuor K, Braun T, Turan JM, Bukusi EA, Nghiem VT. Cost of Home-Based Couples Human Immunodeficiency Virus Counseling and Testing and Human Immunodeficiency Virus Self-Testing During Pregnancy and Postpartum in Southwestern Kenya. Value Health Reg Issues. 2023 Mar;34:125-132. doi: 10.1016/j.vhri.2022.11.003. Epub 2023 Jan 27. PMID 36709657

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In a three-arm randomized controlled trial in southwestern Kenya (2019-2024), we recruited women attending antenatal care, subsequently contacting the male partner.
Pre-assignment Details: A total of 800 pregnant couples (1,600 individuals) were randomized to the home visit intervention (HV, n=267 couples = 534 individuals), HIV self-test kits (HIVST, n=266 couples = 532 individuals), or standard care (SC, n=267 couples = 534 individuals).
Period: Overall Study
Arm/Group | Home Visits | HIV Self-testing | Standard Care
Started | 534 | 532 | 534
Completed | 406 | 424 | 382
Not Completed | 128 | 108 | 152
Not completed — Death | 0 | 1 | 5
Not completed — Adverse Event | 24 | 11 | 13
Not completed — Partner discontinued due to the death of the female participant or adverse event | 24 | 12 | 18
Not completed — Lost to Follow-up | 80 | 84 | 116

BASELINE CHARACTERISTICS:
Population: We recruited 800 couples, 800 females (two-thirds living with HIV at baseline) and 800 male partners. Couples who were eligible and willing, were randomized to either the home-based couple intervention, HIV self-test kits for couples, or the standard care arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Home Visits | HIV Self-testing | Standard Care | Total
Number analyzed (Participants) | 534 | 532 | 534 | 1600
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 267 | 266 | 267 | 800
  Male | 267 | 266 | 267 | 800
Race (NIH/OMB) [Count of Participants; unit: Participants] — All 1600 participants were Blacks from Kenya
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 534 | 532 | 534 | 1600
    White | 0 | 0 | 0 | 0
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — All 1600 participants were non-Hispanics from Kenya
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 534 | 532 | 534 | 1600
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — All participants were from Kenya
  Participants
    Kenya | 534 | 532 | 534 | 1600
Number of couples who had ever tested for HIV as a couple prior to study enrollment [Number; unit: Couples who had ever tested for HIV (=Y)] — Prior couple HIV testing at baseline (all couples), coded as Y=those who had ever tested for HIV as a couple prior to study enrollment, N=those who had never tested for HIV as a couple prior to study enrollment. This is assessed in the questionnaires for all couples regardless of HIV status at baseline. Population: Participants numbers below represent number of couples who had ever tested for HIV as a couple prior to study enrollment (coded as 'Yes' value)
  Couples who had ever tested for HIV (=Y)
    number analyzed (Participants) | 266 | 262 | 262 | 790
    (all) | 105 | 103 | 75 | 283
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 5 | 11 | 21
  Between 18 and 65 years | 529 | 527 | 523 | 1579
  >=65 years | 0 | 0 | 0 | 0
Number of individuals who had ever tested individually for HIV prior to study enrollment [Number; unit: Ever tested for HIV individually (=Y)] — Prior individual HIV testing at baseline as assessed in the questionnaire coded as Y=those who had ever tested for HIV individually prior to study enrollment, N=those who had never tested for HIV individually a prior to study enrollment, completed by all participants at baseline. Population: Number of individuals who had ever tested individually for HIV prior to study enrollment (coded as 'Yes')
  Ever tested for HIV individually (=Y)
    number analyzed (Participants) | 533 | 529 | 531 | 1593
    (all) | 526 | 523 | 517 | 1566
Maternal HIV Viral Suppression (HIV-positive Women) [Count of Participants; unit: Participants] — Viral Load < 200 copies (undetectable) for all HIV-positive women at baseline through medical records. Population: All HIV-positive women at baseline.
  Participants
    number analyzed (Participants) | 118 | 131 | 126 | 375
    (all) | 117 | 124 | 114 | 355

OUTCOME MEASURES:

1. Primary Outcome: Number of Couples Who Tested for HIV as a Couple After Study Enrollment up to 12 Months Postpartum
Description: Number of couples with couple HIV testing uptake during observation period (from baseline to 12 months postpartum), coded as Y=if the couple tested together for HIV up to 12 months postpartum and N=if the couple has not tested together for HIV up to 12 months postpartum. At 3 and 12 months postpartum, each couple member was asked to report whether they had tested together for HIV as a couple at home with HIV self-test kits or at the clinic.
Time Frame: up to 12 months postpartum
Population: Couple HIV Testing and Counseling was defined as testing together with partner at the clinic, home, or with HIV self-test kits at either 3 or 12 months postpartum. Couples with a test at 3 months postpartum only were considered tested.
Measure: Number; unit: Couples tested for HIV as a couple (=Y)
Arm/Group | Home Visits | HIV Self-testing | Standard Care
Number analyzed (Participants) | 203 | 212 | 191
Couples tested for HIV as a couple (=Y) | 114 | 106 | 26
Statistical Analysis 1: Comparison: Home Visits vs Standard Care; Home visits as compared to Standard Care; Test type: Superiority; p < 0.001, Chi-squared; Risk Ratio (RR) = 4.22, 95% CI 2-sided [2.88 to 6.18] — Generalized Estimating Equation model with robust standard errors used. Risk Ratios reported were adjusted for baseline education level, wealth index, length of couple relationship, previous couple testing at baseline, and couple age disparity
Statistical Analysis 2: Comparison: HIV Self-testing vs Standard Care; HIV Self-testing as compared to Standard Care; Test type: Superiority; p < 0.001, Chi-squared; Risk Ratio (RR) = 3.69, 95% CI 2-sided [2.50 to 5.45] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: HIV Re-testing
Description: Re-testing for HIV during pregnancy and postpartum during observation period assessed in the questionnaire.
Time Frame: Up to 12 months postpartum
Population: Individuals HIV Retesting and Counseling was defined as retesting at either 3 or 12 months postpartum after initial baseline testing. Individuals with a retest at 3 months postpartum only were considered to have retested at 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Home Visits | HIV Self-testing | Standard Care
Number analyzed (Participants) | 403 | 416 | 363
Participants | 338 | 367 | 258
Statistical Analysis 1: Comparison: Home Visits vs Standard Care; Comparison of the Home Visit arm with Standard Care; Test type: Superiority; p = .001, Chi-squared; Risk Ratio (RR) = 1.21, 95% CI 2-sided [1.12 to 1.31] — Generalized Estimating Equation model with robust standard errors used. Risk Ratios reported were adjusted for baseline education level, wealth index, length of couple relationship, previous couple testing at baseline, and and couple age disparity
Statistical Analysis 2: Comparison: HIV Self-testing vs Standard Care; Comparison of HIVST arm with Standard Care arm; Test type: Superiority; p = .001, Chi-squared; Risk Ratio (RR) = 1.26, 95% CI 2-sided [1.17 to 1.36] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Number of New Male HIV-positive Diagnoses From Baseline up to 12 Months Postpartum (Intervention Arms Only)
Description: Number of new HIV-positive test results of male partners from baseline to 12 months postpartum and coded as Y=those who had tested for HIV individually up to 12 months postpartum and N=those who had not tested for HIV individually up to 12 months postpartum.
Time Frame: Up to 12 months postpartum
Population: HIV-negative Male Partners at baseline and retained at 12 months postpartum. Data were collected in intervention arms only.
Measure: Number; unit: No. of men with new HIV+ diagnoses (=Y)
Arm/Group | Home Visits | HIV Self-testing | Standard Care
Number analyzed (Participants) | 244 | 256 | 0
No. of men with new HIV+ diagnoses (=Y) | 9 | 2 |

4. Secondary Outcome: Number of New Discordant Couples (Intervention Arms Only)
Description: Number of new HIV serodiscordant couples identified during observation period.
Time Frame: Up to 12 months postpartum
Population: All non-discordant couples at baseline. Data were collected in intervention arms only
Measure: Count of Participants; unit: Participants
Arm/Group | Home Visits | HIV Self-testing | Standard Care
Number analyzed (Participants) | 94 | 98 | 0
Participants | 93 | 35 | 0

5. Secondary Outcome: HIV+ Women Who Utilized All 3 PMTCT Interventions up to 18 Months Postpartum
Description: Composite variable based on self-report data from women's questionnaires, coded as Y=those who were coded as Y on the three variables described below and N= those who were coded as N on one, two, or three variables described below: (1) mothers use of antiretrovirals (ARVs) (Y=those mothers who have used ARVs from baseline up to 18 months postpartum/N=those mothers who have not used ARVs at any time point between baseline up to 18 months postpartum), (2) prophylactic ARVs given to the infant (Y=those infants who were given prophylactic ARVs up to 18 months after the birth/N=those infants who were not given prophylactic ARVs at any point from birth up to 18 months after the birth), and (3) Y=if exclusive breastfeeding was practiced up to 6 months after the birth and N=if exclusive breastfeeding was not practiced up to 6 months after the birth.
Time Frame: Up to 18 months postpartum
Population: HIV positive women retained up to 18-months follow-up
Measure: Number; unit: HIV+ women w/all 3 PMTCT interventions
Arm/Group | Home Visits | HIV Self-testing | Standard Care
Number analyzed (Participants) | 107 | 98 | 89
HIV+ women w/all 3 PMTCT interventions | 31 | 28 | 28

6. Secondary Outcome: Women Who Utilized All 4 MCH Services up to 3 Months Postpartum
Description: Composite variable based on self-report data from women's questionnaires: Y=if all described variables coded as Y, N=if at least one of the following variables coded as N: (1) Y=if a woman completed at least four antenatal care (ANC) visits during this pregnancy, N=if a woman completed less than four ANC visits during this pregnancy; (2) Y=if a childbirth was with a skilled attendant, N=if a childbirth was not with a skilled attendant; (3) Y=if a postpartum check-up was completed for a woman and N=if the women did not have a postpartum check-up, and (4) Y=if the infant had a postnatal check-up, N=if a if a postnatal check-up was not completed for the infant. These are assessed in the follow-up questionnaires completed up to 3 months postpartum.
Time Frame: Up to 3 months postpartum
Population: Women retained up to 3 months postpartum
Measure: Number; unit: Women who utilized all 4 MCH services
Arm/Group | Home Visits | HIV Self-testing | Standard Care
Number analyzed (Participants) | 188 | 190 | 172
Women who utilized all 4 MCH services | 116 | 103 | 91

7. Secondary Outcome: Pre-Exposure Prophylaxis (PrEP) Uptake (HIV Negative at Baseline)
Description: Initiation of PrEP by participants with HIV-negative status at baseline, assessed at each follow-up in the questionnaires up to 18 months after the baby's birth.
Time Frame: Up to 18 months postpartum
Population: HIV negative participants at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Home Visits | HIV Self-testing | Standard Care
Number analyzed (Participants) | 369 | 399 | 348
Participants | 47 | 49 | 46

8. Secondary Outcome: Number of HIV-positive Women Not Linked to HIV Care at Baseline Reported Being Linked to HIV Care at 12 Months Postpartum
Description: Number of HIV-positive women not linked to HIV care at baseline reported being linked to HIV care at 12 months postpartum assessed at baseline and in the follow-up questionnaires completed up to 12 months postpartum and confirmed through medical records. Coded as Y=if HIV-positive woman at baseline and not linked to HIV care at baseline reported being linked to HIV care at 12 months postpartum. Coded as N=if HIV-positive woman at baseline and not linked to HIV care at baseline reported not being linked to HIV care at 12 months postpartum.
Time Frame: Up to 12 months postpartum
Population: Number of HIV-positive women not linked to HIV care at baseline reported being linked to HIV care at 12 months postpartum (coded as "yes")
Measure: Number; unit: Number of women linked to HIV care(=Y)
Arm/Group | Home Visits | HIV Self-testing | Standard Care
Number analyzed (Participants) | 4 | 1 | 2
Number of women linked to HIV care(=Y) | 4 [0 to 0] | 1 [0 to 22.9] | 1 [0 to 3.3]

9. Secondary Outcome: Number of HIV-positive Women at Baseline Retained in HIV Care up to 12 Months Follow-up
Description: Woman's retention in HIV care assessed for HIV-positive women at baseline and in the follow-up questionnaires completed up to 12 months postpartum and confirmed through medical records. Coded as Y=if HIV-positive woman at baseline was retained in HIV care up to 12 months postpartum and N=if HIV-positive woman at baseline has not been retained in HIV up to 12 months postpartum.
Time Frame: Up to 12 months postpartum
Population: Number of HIV-positive women at baseline retained in HIV care up to 12-months follow-up (coded as "Yes')
Measure: Number; unit: Number of women retained in HIV care(=Y)
Arm/Group | Home Visits | HIV Self-testing | Standard Care
Number analyzed (Participants) | 151 | 165 | 160
Number of women retained in HIV care(=Y) | 151 | 165 | 159

10. Secondary Outcome: Mean Woman's Adherence to HIV Treatment (ART) (HIV-positive Women Retained up to 12-months Follow-up)
Description: Mean self-reported adherence to ART was assessed using self-report questionnaire data for HIV-positive women at baseline and in the follow-up questionnaires completed up to 12 months postpartum. Adherence was measured using a 3-item adherence scale (Wilson et al., 2014) with items on number of missed doses, self-evaluation of how good a job she was doing with adherence, and how often taken as recommended; all for the last 30 days. An adherence score (possible range 0-100%) was calculated for each woman at each time point.
Time Frame: Up to 12 months postpartum
Population: HIV-positive women retained up to 12-months follow-up
Measure: Mean (Standard Deviation); unit: Adherence score
Arm/Group | Home Visits | HIV Self-testing | Standard Care
Number analyzed (Participants) | 151 | 165 | 160
Adherence score | 73.9 (7.5) | 71.8 (7.4) | 71.3 (8.8)

11. Secondary Outcome: Mean Number of HIV Care Visits (HIV-positive Women Retained up to 12-months Follow-up)
Description: Mean number of HIV care visits assessed for HIV-positive women at baseline and in the follow-up questionnaires completed up to 12 months postpartum and confirmed through medical records.
Time Frame: Up to 12 months postpartum
Population: HIV-positive women retained up to 12-months follow-up
Measure: Mean (Standard Deviation); unit: Number of visits
Arm/Group | Home Visits | HIV Self-testing | Standard Care
Number analyzed (Participants) | 151 | 165 | 160
Number of visits | 4.7 (1.3) | 4.7 (1.4) | 4.7 (1.3)

12. Secondary Outcome: Number of HIV-positive Men Not Linked to HIV Care at Baseline Reported Being Linked to HIV Care at 12 Months Postpartum
Description: Number of HIV-positive men not linked to HIV care at baseline reported being linked to HIV care at 12 months postpartum assessed at baseline and in the follow-up questionnaires completed up to 12 months postpartum and confirmed through medical records. Coded as Y=if HIV-positive man at baseline and not linked to HIV care at baseline reported being linked to HIV care at 12 months postpartum. Coded as N=if HIV-positive man at baseline and not linked to HIV care at baseline reported not being linked to HIV care at 12 months postpartum.
Time Frame: Up to 12 months postpartum
Population: Number of HIV-positive men not linked to HIV care at baseline reported being linked to HIV care at 12 months postpartum (coded as "yes")
Measure: Number; unit: Number of men linked to HIV care (=Y)
Arm/Group | Home Visits | HIV Self-testing | Standard Care
Number analyzed (Participants) | 2 | 1 | 0
Number of men linked to HIV care (=Y) | 2 | 1 |

13. Secondary Outcome: Number of HIV-positive Men at Baseline Retained in HIV Care up to 12 Months Follow-up
Description: Men's retention in HIV care assessed for HIV-positive men at baseline and in the follow-up questionnaires completed up to 12 months postpartum and confirmed through medical records. Coded as Y=if HIV-positive man at baseline was retained in HIV care up to 12 months postpartum and N=if HIV-positive man at baseline has not been retained in HIV up to 12 months postpartum.
Time Frame: Up to 12 months postpartum
Population: Number of HIV-positive men at baseline retained in HIV care up to 12-months follow-up (coded as "Yes')
Measure: Number; unit: Number of men retained in HIV care(=Y)
Arm/Group | Home Visits | HIV Self-testing | Standard Care
Number analyzed (Participants) | 14 | 6 | 17
Number of men retained in HIV care(=Y) | 14 | 6 | 17

14. Secondary Outcome: Mean Man's Adherence to HIV Treatment (ART) (HIV-positive Men Retained up to 12 Months Postpartum)
Description: Mean self-reported adherence to ART assessed for HIV-positive men at baseline and in the follow-up questionnaires completed up to 12 months postpartum and confirmed through medical records. Mean self-reported adherence to ART was assessed using self-report questionnaire data for HIV-positive men at baseline and in the follow-up questionnaires completed up to 12 months postpartum. Adherence was measured using a 3-item adherence scale (Wilson et al., 2014) with items on number of missed doses, self-evaluation of how good a job he was doing with adherence, and how often taken as recommended; all for the last 30 days. An adherence score (possible range 0-100%) was calculated for each male partner at each time point using these three items.
Time Frame: Up to 12 months postpartum
Population: HIV-positive men retained up to 12 months postpartum.
Measure: Mean (Standard Deviation); unit: Adherence score
Arm/Group | Home Visits | HIV Self-testing | Standard Care
Number analyzed (Participants) | 13 | 26 | 39
Adherence score | 70.7 (7.9) | 66 (7.9) | 65 (8.2)

15. Secondary Outcome: Mean Number of HIV Care Visits (HIV-positive Men Retained up to 12 Months Postpartum)
Description: Mean number of HIV care visits assessed for HIV-positive men from baseline up to 12 months postpartum.
Time Frame: Up to 12 months postpartum
Population: HIV-positive men retained up to 12 months postpartum
Measure: Mean (Standard Deviation); unit: Number of visits
Arm/Group | Home Visits | HIV Self-testing | Standard Care
Number analyzed (Participants) | 13 | 26 | 39
Number of visits | 3.2 (1.2) | 2.4 (0.7) | 2.9 (1.5)

16. Secondary Outcome: Maternal HIV Viral Suppression (HIV-positive Women Retained up to 18-months Follow-up)
Description: Viral Load < 200 copies (undetectable) for all HIV-positive women at baseline and 18 months postpartum through medical records.
Time Frame: Up to 18 months postpartum
Population: Women living with HIV at initial baseline testing and retained at 18-month follow-up Viral load (VL) testing done in late pregnancy or 3 months, 12, and 18 months postpartum.
  Analysis included those with at least one follow up VL measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Home Visits | HIV Self-testing | Standard Care
Number analyzed (Participants) | 118 | 131 | 126
Participants | 117 | 124 | 114
Statistical Analysis 1: Comparison: Home Visits vs Standard Care; Comparison of the Home Visit arm with Standard Care; Test type: Superiority; p = .011, Chi-squared; Risk Ratio (RR) = 1.08, 95% CI 2-sided [1.03 to 1.12] — Generalized Estimating Equation model (binomial family and log link) with robust standard errors used. Risk Ratios reported were adjusted for baseline education level, wealth, length of couple relationship, and couple age disparity
Statistical Analysis 2: Comparison: HIV Self-testing vs Standard Care; Comparison of the HIVST arm with Standard Care; Test type: Superiority; p = 0.011, Chi-squared; Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.97 to 1.08] — [estimate comment as in outcome 16, analysis 1]

17. Secondary Outcome: HIV-free Child Survival
Description: Child alive and HIV-free at 18 months after the birth. This is assessed in a brief interview and confirmed through medical records.
Time Frame: 18 months after the birth
Population: Infants with 18 month final HIV testing and survival outcome. No stillbirths or miscarriages included in denominator.
Measure: Count of Participants; unit: Participants
Arm/Group | Home Visits | HIV Self-testing | Standard Care
Number analyzed (Participants) | 141 | 146 | 146
Participants | 130 | 141 | 142
Statistical Analysis 1: Comparison: Home Visits; Test type: Other; p = 0.087, Log Rank; Kaplan Meier estimates = 0.92, 95% CI 2-sided [0.86 to 0.95]
Statistical Analysis 2: Comparison: HIV Self-testing; Test type: Other; p = 0.087, Log Rank; Kaplan Meier estimates = 0.96, 95% CI 2-sided [0.91 to 0.98]
Statistical Analysis 3: Comparison: Standard Care; Test type: Other; p = 0.087, Log Rank; Kaplan Meier estimates = 0.98, 95% CI 2-sided [0.93 to 0.99]

18. Secondary Outcome: Number of Infants of HIV-positive Mothers Who Tested HIV+ up to 18 Months Postpartum
Description: Number of infants of HIV-positive mothers who tested HIV+ up to 18 months postpartum based on medical records. This is be a Y/N variable with Y if the infant tested HIV+ up to 18 months postpartum and N if they did not test HIV+.
Time Frame: Up to 18 months after birth
Population: Number of infants of HIV-positive women retained up to 18-months follow-up (coded as 'Yes')
Measure: Number; unit: Infants of HIV+ mothers who tested HIV+
Arm/Group | Home Visits | HIV Self-testing | Standard Care
Number analyzed (Participants) | 133 | 142 | 144
Infants of HIV+ mothers who tested HIV+ | 1 | 1 | 0

19. Secondary Outcome: Time to First Infant HIV Test (Infants of HIV-positive Women Retained up to 18-months Follow-up)
Description: Time to first infant HIV test based on medical records. This is the number of weeks since the baby's birth to the first HIV test and is reported as a median weeks value for each study arm.
Time Frame: Up to 18 months after birth
Population: Infants of HIV-positive women retained up to 18-months follow-up.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Home Visits | HIV Self-testing | Standard Care
Number analyzed (Participants) | 141 | 146 | 146
Weeks | 6.6 [6 to 10] | 6.3 [6 to 8.6] | 6.3 [6 to 8.2]

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up: up to 18 months postpartum
Description: Adverse events were self-reported, reported during regular follow-ups, or detected through data abstraction from medical records. Reporting followed standard operating procedures, guidance from ethical boards and funder, as well as the study Data Safety Monitoring Board process review and reporting. Couples who experienced adverse pregnancy outcomes were discontinued from the study as the intervention sessions focused on health during pregnancy and postpartum.
Arm/Group | Home Visits | HIV Self-testing | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/534 | 1/532 | 5/534
Serious Adverse Events (participants affected / at risk) | 24/534 | 11/532 | 13/534
Other Adverse Events (participants affected / at risk) | 11/534 | 21/532 | 12/534
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home Visits (N=534) | HIV Self-testing (N=532) | Standard Care (N=534)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 2 (2) — Loss of fetus before 28 weeks gestation
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 3 (3) | 6 (6) — No signs of life at birth > 28 weeks gestation
Neonatal Deaths (Pregnancy, puerperium and perinatal conditions) | 11 (11) | 1 (1) | 4 (4) — Death in the first 28 days of life
Infant Deaths (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 4 (4) | 1 (1) — Death between 1 month to <1 year of age
Child death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) — Death ≥1 year of age
Hospitalization (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) — Hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home Visits (N=534) | HIV Self-testing (N=532) | Standard Care (N=534)
Separation/relationship dissolution (Social circumstances) | 2 (2) | 10 (10) | 2 (2) — Couples move out of home or relationship dissolution
New intimate partner violence (Social circumstances) | 6 (6) | 10 (10) | 8 (8) — Intimate Partner Violence (physical and/or sexual)
Depression (Psychiatric disorders) | 3 (3) | 1 (1) | 2 (2) — Score ≥ 10 points on the PHQ-8 scale

LIMITATIONS AND CAVEATS:
Investigators enrolled a selected sample of couples who were living together in stable relationships with both partners of the couple willing to participate in the research. The study used self-report measures for the primary outcome of CHTC for the comparison groups and several of the intermediate variables, which may be subject to recall and other reporting biases. Another limitation was introduced by the occurrence of the COVID-19 pandemic in the middle of the study period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/39/NCT03547739/Prot_SAP_ICF_000.pdf